CLINICAL TRIAL: NCT04490434
Title: A Randomized, Open-label, Multiple-dose Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetic Drug-drug Interaction Between DWP14012 and Three Different Kinds of NSAIDs in Healthy Male Volunteers
Brief Title: Drug-drug Interaction Between DWP14012 and Three Different Kinds of NSAIDs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DW_DWP14012005
Record Dates: First submitted 2020-04-24; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — fexuprazan; Celecoxib; Naproxen; Meloxicam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1, A (DWP14012/Celecoxib) (Experimental): Patients treated with DWP14012, Celecoxib will be enrolled. DDI will be evaluated.
  Interventions: Drug: DWP14012; Drug: Celecoxib
- Cohort 1, B (DWP14012/Celecoxib) (Experimental): Patients treated with DWP14012, Celecoxib will be enrolled. DDI will be evaluated.
  Interventions: Drug: DWP14012; Drug: Celecoxib
- Cohort 2, C (DWP14012/Naproxen) (Experimental): Patients treated with DWP14012, Naproxen will be enrolled. DDI will be evaluated.
  Interventions: Drug: DWP14012; Drug: Naproxen
- Cohort 2, D (DWP14012/Naproxen) (Experimental): Patients treated with DWP14012, Naproxen will be enrolled. DDI will be evaluated.
  Interventions: Drug: DWP14012; Drug: Naproxen
- Cohort 3, E (DWP14012/Meloxicam) (Experimental): Patients treated with DWP14012, Meloxicam will be enrolled. DDI will be evaluated.
  Interventions: Drug: DWP14012; Drug: Meloxicam
- Cohort 3, F (DWP14012/Meloxicam) (Experimental): Patients treated with DWP14012, Meloxicam will be enrolled. DDI will be evaluated.
  Interventions: Drug: DWP14012; Drug: Meloxicam

INTERVENTIONS:
Drug: DWP14012 — DWP14012 40mg, bid
Drug: Celecoxib — Celecoxib 200mg, bid
  Arms: Cohort 1, A (DWP14012/Celecoxib); Cohort 1, B (DWP14012/Celecoxib)
Drug: Naproxen — Naproxen 500mg, bid
  Arms: Cohort 2, C (DWP14012/Naproxen); Cohort 2, D (DWP14012/Naproxen)
Drug: Meloxicam — Meloxicam 15mg, qd
  Arms: Cohort 3, E (DWP14012/Meloxicam); Cohort 3, F (DWP14012/Meloxicam)

SUMMARY:
drug-drug interaction between DWP14012 and three different kinds of NSAIDs

DETAILED DESCRIPTION:
to evaluate the safety/tolerability and pharmacokinetic drug-drug interaction between DWP14012 and three different kinds of NSAIDs in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult Caucasian or Japanese or Korean aged 19 to 50 (inclusive) years, at the time of screening.
* Subjects weighing between 50 kg and 90 kg with BMI between 18 and 27 kg/m2 (inclusive) at screening visit.

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Those who have gastrointestinal diseases or past history of gastrointestinal diseases (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux, Crohn's disease etc.) that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple appendectomy and herniotomy)
* Those whose plasma AST (SGOT) and ALT (SGPT) exceed 1.5 times to the upper limit of the normal range in screening including additional examinations prior to randomization
* Subjects who have participated and taken investigational drug in any other clinical trial (including bioequivalence study) within six months prior to study drug administration
* Subjects who have donated a unit of whole blood within two months or blood components within one month prior to study drug administration

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Arm A, Cmax,ss of Celecoxib | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Maximum measured plasma concentration at steady-state
Arm A, AUCτ,ss of Celecoxib | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Area under the plasma concentration-time curve
Arm B, Cmax,ss of DWP14012 | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Maximum measured plasma concentration at steady-state
Arm B, AUCτ,ss of DWP14012 | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Area under the plasma concentration-time curve
Arm C, Cmax,ss of Naproxen | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Maximum measured plasma concentration at steady-state
Arm C, AUCτ,ss of Naproxen | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Area under the plasma concentration-time curve
Arm D, Cmax,ss of DWP14012 | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Maximum measured plasma concentration at steady-state
Arm D, AUCτ,ss of DWP14012 | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 11,(0 hours (pre-dose), 0.5~48 hours)
  Area under the plasma concentration-time curve
Arm E, Cmax,ss of Meloxicam | Day 7,(0 hours (pre-dose), 1~72 hours) / Day 16,(0 hours (pre-dose), 1~72 hours)
  Maximum measured plasma concentration at steady-state
Arm E, AUCτ,ss of Meloxicam | Day 7,(0 hours (pre-dose), 1~72 hours) / Day 16,(0 hours (pre-dose), 1~72 hours)
  Area under the plasma concentration-time curve
Arm D, Cmax,ss of DWP14012 | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 13,(0 hours (pre-dose), 0.5~48 hours)
  Maximum measured plasma concentration at steady-state
Arm D, AUCτ,ss of DWP14012 | Day 5,(0 hours (pre-dose), 0.5~48 hours) / Day 13,(0 hours (pre-dose), 0.5~48 hours)
  Area under the plasma concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Jang In-Jin, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Won H, Kim E, Chae J, Lee H, Cho JY, Jang IJ, Chung JY, Kim MG, Lee S. Pharmacokinetic interactions between fexuprazan, a potassium-competitive acid blocker, and nonsteroidal anti-inflammatory drugs in healthy males. Clin Transl Sci. 2024 May;17(5):e13798. doi: 10.1111/cts.13798. PMID 38700290